CLINICAL TRIAL: NCT03610841
Title: Evaluation of the Possible Relationship Between Preterm Labor and Periodontal Disease With Clinical Periodontal, Biochemical and Microbiological Data
Brief Title: Evaluation of the Possible Relationship Between Periodontal Disease and Preterm Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Gul Yildiz Telatar, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 40465587-26
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Preterm Labor; Periodontal Disease
MeSH Terms: conditions — Obstetric Labor, Premature; Periodontal Diseases | interventions — Blood Specimen Collection; Urinalysis; Diet, Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples from four centers will be taken from the maternal and fetal surfaces of the placenta Saliva samples of pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm labor: Workgroup consists of patients which diagnosed with preterm labor between the age of 21 and 34
  Interventions: Diagnostic Test: preterm labor; Diagnostic Test: healthy
- healthy: 24-36 6/7 weeks of pregnant between the age of 21 and 34
  Interventions: Diagnostic Test: preterm labor; Diagnostic Test: healthy

INTERVENTIONS:
Diagnostic Test: preterm labor — liver function tests, kidney function tests and platelets measures the ratio of protein to creatinine
  Other Names: blood sample, urine test
Diagnostic Test: healthy — liver function tests, kidney function tests and platelets measures the ratio of protein to creatinine
  Other Names: blood sample, urine test

SUMMARY:
The primary objective of the study is to assess the incidence and severity of the periodontal infection of patients with preterm labor.

The secondary objective of the study is to analyze the relationship between preterm labor and periodontal infection, using clinical, biochemical and microbiological methods.

DETAILED DESCRIPTION:
Preterm infants are born prior to completion of 37 weeks of gestation. Periodontal disease is a subclinical and persistent infection source which induces the systemic inflammatory reactions and increases the risk of preterm labor. It is believed that the results will set light to the etiology of preterm labor and will help to develop strategies to prevent the disease.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preterm labor
* 37. weeks of pregnant women with no history of preterm labor

Exclusion Criteria:

* Genitourinary infection
* pregnancy or pre-pregnancy hypertension
* HIV infection
* diabetes mellitus
* multiple pregnancy, preterm labor / low birth weight
* smoker and alcohol use history
* IVF pregnancy
* placental, cervical and uterine anomalies
* pregnancy with intrauterine growth retardation
* pregnancies with congenital or chromosomal fetal anomalies
* significant vaginal bleeding
* infertility stories
* drug addicts
* poor socioeconomic level

Ages: 21 Years to 34 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: The study is planned to be a case-control study. Workgroup consists of 50 patients which diagnosed with preterm labor between the age of 21 and 34. Control group consists of healthy females 24-36 6/7 weeks of pregnant with no history of preterm labor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-17 (Actual); Primary Completion 2018-09-17 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
prostaglandin E2 | 1 Day
  prostaglandin E2 levels will be evaluated in salivary, serum and placenta samples using ELISA test Normal value:29-97 pg / ml
TNF-Alpha | 1 day
  TNF-Alpha levels will be evaluated in salivary, serum and placenta samples using ELISA test Normal value:42-203pg/ml
IL-1beta | 1 day
  IL-1beta levels will be evaluated in salivary, serum and placenta samples using ELISA test Normal value:3-227pg/ml

SECONDARY OUTCOMES:
Porphyromonas gingivalis | 1 Day
  Presence of Porphyromonas gingivalis will be checked by rPCR method. Score 1: Present Score 2: None
Tannerella Forsythia | 1 Day
  Presence of Tannerella Forsythia will be checked by rPCR method. Score:1 Present. Score 2: None

CONTACTS AND LOCATIONS:
Locations (6):
- Turkey (Türkiye) (5):
  - Ege University Dentistry Faculty, Izmir
  - İzmir Health Sciences University, Tepecik Training and Research Hospital Department of Obstetrics and Gynecology, Izmir
  - Recep Tayyip Erdogan University Dentistry Faculty, Rize
  - Recep Tayyip Erdogan University Faculty of Medicine, Rize
  - Recep Tayyip Erdogan University, Rize
- Glaskow Dental School , School of Medicine University of Glasgow, Glaskow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be available within 6 months of study completion

REFERENCES:
- [Background] Puertas A, Magan-Fernandez A, Blanc V, Revelles L, O'Valle F, Pozo E, Leon R, Mesa F. Association of periodontitis with preterm birth and low birth weight: a comprehensive review. J Matern Fetal Neonatal Med. 2018 Mar;31(5):597-602. doi: 10.1080/14767058.2017.1293023. Epub 2017 Feb 28. PMID 28282773
- See also: Association of periodontitis with preterm birth and low birth weight — http://www.ncbi.nlm.nih.gov/pubmed/28282773